CLINICAL TRIAL: NCT01637350
Title: The Effect of Blood Glucose to Different Digestive Tract Reconstruction After Gastrectomy of Gastric Cancer With Type 2 Diabetes
Brief Title: Digestive Tract Reconstruction After Gastrectomy of Gastric Cancer With Type 2 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CIH-WXN-201205001
Record Dates: First submitted 2012-07-06; First posted 2012-07-11 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2012-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Subtotal gastrectomy , BillrothⅠ
  Interventions: Procedure: digestive tract reconstruction
- Subtotal gastrectomy , BillrothⅡ
  Interventions: Procedure: digestive tract reconstruction
- total gastrectomy, jejunal interposition
  Interventions: Procedure: digestive tract reconstruction
- total gastrectomy , Roux-en-Y
  Interventions: Procedure: digestive tract reconstruction

INTERVENTIONS:
Procedure: digestive tract reconstruction — Subtotal gastrectomy with BillrothⅠ or BillrothⅡ, total gastrectomy with jejunal interposition or Roux-en-Y reconstruction
  Other Names: no other names

SUMMARY:
Different digestive tract reconstruction will affect the blood glucose level of gastric cancer with type 2 diabetes. Subtotal gastrectomy with Billroth II reconstruction and total gastrectomy with Roux-en-Y reconstruction may help to improve glycaemic control which includes fasting blood glucose, postprandial blood glucose, glycosylated hemoglobin, C -peptide and body weight of gastric cancer patients with type 2 diabetes.

DETAILED DESCRIPTION:
Different digestive tract reconstruction will affect the blood glucose level of gastric cancer with type 2 diabetes. Subtotal gastrectomy with Billroth II reconstruction and total gastrectomy with Roux-en-Y reconstruction may help to improve glycaemic control which includes fasting blood glucose, postprandial blood glucose, glycosylated hemoglobin, C -peptide and body weight of gastric cancer patients with type 2 diabetes.

The investigators will observed fasting blood glucose, postprandial blood glucose, glycosylated hemoglobin, C -peptide and body weight of the patients preoperation, 14 days postoperation 3 month and 6month postoperation. The investigators will observed the effect of blood glucose to different digestive tract reconstruction after gastrectomy of gastric cancer with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old,gastric cancer ,can be performed operation
2. with type 2 diabetes,fasting blood glucose > 6.1mmol/L
3. without serious underlying diseases which may affect the metabolism and nutrient uptake
4. without serious underlying diseases which may affect anesthesia and operation
5. can be performed subtotal or total gastrectomy, predicted survival period > 6months
6. no other abdominal operation
7. preoperation consultation
8. informed consent

Exclusion Criteria:

1. recurrent,metastasis or die
2. patient requests for quit
3. pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: gastric cancer with type 2 diabetes,18~75 years old,without serious underlying diseases
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Yan, Doctor, Study Director — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China